CLINICAL TRIAL: NCT06930521
Title: JUdicious Surveillance for Trastuzumab Induced Cardiotoxicity in the First Year (JUSTIFY): a Randomized Controlled Trial
Brief Title: JUdicious Surveillance for Trastuzumab Induced Cardiotoxicity in the First Year
Acronym: JUSTIFY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Husam Abdel-Qadir, Cardiologist, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 5034
Record Dates: First submitted 2025-03-31; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Health; Breast Cancer; Breast Cancer Early Stage Breast Cancer (Stage 1-3); Cardio-oncology; Circulatory and Respiratory Health; Clinical and Translational Cardiovascular Sciences; Health Services and Systems - Healthcare Effectiveness &Amp; Outcomes
Keywords: Trastuzumab; Cardiac imaging; Her-2 positive breast cancer; Echocardiography; Cardiotoxicity; Left ventricular ejection fraction; Heart failure; Randomized controlled trial; Nuclear imaging; Non-inferiority
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Heart Failure

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups with regards to the frequency of mandatory echocardiograms:
  Group 1 - Standard of Care Group: Participants in this group will receive imaging before cycles 1, 5, 9, and 13 of trastuzumab (or every 3 months) and another echocardiogram after completion of trastuzumab (within 100 days after completion of HER2TT).
  Group 2 - Judicious Imaging Group: This group will get less echocardiograms based on their risk of developing heart failure. People who do not have any issues that predispose to heart failure are categorized as low risk and will get an echocardiogram once every 6 months. People who have factors that may predispose to heart failure are categorized as intermediate risk and will get an echocardiogram approximately once every 4 months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): The SOC arm will receive imaging before cycles 1, 5, 9, and 13 (in keeping with the FDA product label), then at the end of HER2-TT, i.e., imaging every 3 months for uninterrupted adjuvant HER2TT.
- Judicious Imaging (Experimental): This group will get less echocardiograms based on their risk of developing heart failure. People who do not have any issues that predispose to heart failure are categorized as low risk and will get an echocardiogram once every 6 months. People who have factors that may predispose to heart failure are categorized as intermediate risk and will get an echocardiogram approximately once every 4 months.
  Interventions: Diagnostic Test: Intervention - Low Risk Group OR Intermediate Risk Group

INTERVENTIONS:
Diagnostic Test: Intervention - Low Risk Group OR Intermediate Risk Group — Participants will be randomized to judicious imaging (decreased imaging frequency based on HF risk category) or SOC (imaging every 3 months). Participants who do not have any HF risk factors will be categorized as low risk, while participants with at least one risk factor will be categorized as intermediate risk for HF.
  Low Risk (zero risk factors): imaging before cycles 1 and 9 of HER2-TT (i.e., at baseline and near the halfway mark, corresponding to 2 fewer studies than SOC in Year 1), then after the end of HER2TT. This translates to imaging every 6 months for uninterrupted adjuvant HER2TT.
  Intermediate Risk (any risk factors): imaging before cycles 1, 6, and 12 of HER2-TT (i.e., at baseline and near the 1/3 and 2/3 marks, corresponding to 1 fewer study than SOC in Year 1), then at end of HER2TT. This translates to imaging every 4 months for uninterrupted adjuvant HER2TT.
  Arms: Judicious Imaging

SUMMARY:
This study focuses on male and female patients being treated for breast cancer that is positive for the HER2 receptor which requires special treatments targeting that receptor. The problem is that these treatments, while effective for the cancer, can sometimes harm the heart. Because of this, patients have to undergo heart tests every three months during treatment, even if they have no history of heart disease or feel fine.

The guidelines for these regular heart tests were established decades ago when these treatments were first introduced, but research shows that most of these tests don't actually change the treatment plan. This suggests that many patients are going through unnecessary tests, which can cause stress, delay treatments, and increase healthcare costs.

To address this, the researchers propose a new study with 300 patients with HER2 positive breast cancer to test a more personalized approach to cardiac surveillance. Participants will be classified based on their risk of heart problems: low or intermediate. Instead of testing every patient every three months, those in the intermediate group will be tested every 4 months, and those in the low-risk group will be tested every 6 months. The researchers will compare this new approach to the current system to see if fewer tests are just as safe and effective.

The researchers will measure heart health, how well cancer treatments are completed, and how patients feel about having fewer tests. If this new approach works, it could save money and reduce the burden on female patients without risking their health.

ELIGIBILITY:
Inclusion Criteria:

1. Stage 1-3 breast cancer (BC).
2. Age 18-79 years.
3. HER-2 positive BC with planned HER2 targeted therapy (HER2TT) for curative intent.

Exclusion Criteria:

1. Distant metastases detected clinically, radiographically, or histologically
2. Baseline echocardiogram images of insufficient quality for a quantitative assessment of left ventricular ejection fraction (LVEF)
3. Pre-existing cardiovascular disease, defined as:

   1. Prior myocardial infarction (even if LVEF has normalized)
   2. Prior heart failure (HF, including patients with preserved ejection fraction and normalized LVEF)
   3. Baseline LVEF <55%
   4. Atrial fibrillation
   5. Greater than moderate valvular disease (i.e., severe, or moderate-severe)
4. Cumulative anthracycline exposure ≥250mg/m2 before starting HER2TT
5. New York Heart Association Functional Class II, III or IV, or Eastern Cooperative Oncology Group score >2*
6. Symptoms potentially due to serious cardiac disease as per investigator's judgement* *Exclusion criterion adopted as they make clinical assessment less reliable to detect emergent HF.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite endpoint encompassing heart health, patient well-being, treatment completion, and imaging frequency in combination, while assessing priority to more important measures. | From enrollment to the end of treatment at 48 weeks
  The primary outcome is a hierarchical composite endpoint for patients with BC receiving HER2-targeted therapy (HER2TT). Participant in the intervention group is compared to participants in the control group based on the following outcomes, in order:
  1. Clinically overt heart failure (determined as a binary event Y/N, per standardized definition)
  2. Premature discontinuation of HER2TT (determined as a binary event Y/N, per clinical records)
  3. Patient-reported outcome measures (PROM) of anxiety/depression, stress and treatment burden: desirable outcome is a better scores in ≥2 of 3 PROMs-Treatment Burden Questionnaire, Hospital Anxiety and Depression Scale, Perceived Stress Scale
  4. Asymptomatic cardiotoxicity at end of HER2TT (per criteria, based on LVEF change from baseline to 12 months echocardiograms)
  5. Time to complete HER2TT (shorter is better)-number of weeks between 1st and last HER2TT
  6. Total cardiac imaging tests during HER2TT (fewer is better)-total assessments of LVEF

CONTACTS AND LOCATIONS:
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No